CLINICAL TRIAL: NCT03558529
Title: ExPRESS:2 (Experiences of Psychosis Relapse: Early Subjective Signs) Longitudinal Feasibility Study
Brief Title: Feasibility and Acceptability of a Smartphone App to Assess Early Warning Signs of Psychosis Relapse
Acronym: ExPRESS:2
Status: Completed | Type: Observational
Sponsor: Manchester Academic Health Science Centre (Other)
Responsible Party: Principal Investigator, Emily Eisner, Principal Investigator, Manchester Academic Health Science Centre
Other Study IDs: 157360; MR/J500410/1 (Other Grant/Funding Number: Medical Research Council); MR/K500823/1 (Other Grant/Funding Number: Medical Research Council); MR/K501311/1 (Other Grant/Funding Number: Medical Research Council)
Record Dates: First submitted 2018-05-22; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Schizophrenia Relapse; Schizophrenia; Schizo Affective Disorder; Psychotic Disorders; Psychosis
Keywords: relapse; early signs; basic symptoms; smartphone app; mhealth
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
About 1 in 100 people will experience an episode of psychosis. Some people will only experience one 'psychotic episode' and about a quarter of people make a full recovery. Others will have recurring periods of problems ('relapses'), perhaps at times of particular stress. As people often find psychosis distressing, this study looks at ways to help them stay well in the future.

There is growing evidence that 'early signs' interventions can prevent relapses of psychosis. Early signs are things that might happen when people start to become unwell. For example some people start to sleep badly when they are becoming unwell. Most people with psychosis can identify early signs emerging in the weeks before relapse. In early signs interventions, service users are taught to recognise early signs that their mental health may be deteriorating so that they can take action to avoid becoming unwell.

Although early signs interventions show promise, the investigators suggest that they can be improved by more accurate assessment of relapse risk. This might be achieved by monitoring 'basic symptoms' in addition to conventional early signs of relapse. Basic symptoms are subtle, subclinical disturbances in one's experience of oneself and the world. Typical basic symptoms include: changes in perceptions, such as increased vividness of colour vision; impaired tolerance to certain stressors; difficulty finding or understanding common words.

In this study the investigators want to design and test a mobile phone app to help monitor basic symptoms. They hope that the app might help service users to stay well in the future. During the study the investigators will ask participants to use the app once a week for 6 months. At the end of the study they will interview them about their experiences of using the phone app and participating in the study.

DETAILED DESCRIPTION:
BACKGROUND

Around 80% of those treated for a first episode of psychosis relapse within five years, with cumulative relapse rates of 78% and 86% for second and third relapses during this period. Relapses can be devastating for the individual and their family, may lead to a deteriorating course of illness and frequently require hospital admission, the principal source of schizophrenia's annual direct cost to the NHS of over £3.9 billion. Given the prevalence and considerable negative consequences of relapse, it is clear that relapse prevention strategies for those with psychosis are a priority.

There is growing evidence that interventions monitoring 'early signs' can be effective in preventing relapses of psychosis. Such interventions work on the premise that timely prediction of relapses will allow preventative action to be taken, minimizing the chance of full relapse occurring. The patient is assisted in identifying and monitoring early signs of relapse, and in developing concrete action plans for dealing with them (e.g. short term medication increases, stress reduction techniques, intensive psychological support). Early signs reported to emerge in the weeks before a relapse include: anxiety, dysphoria, insomnia, poor concentration, attenuated psychotic symptoms (Early Signs Scale, ESS) and fear of relapse (Fear of Recurrence Scale, FoRSe). However, such checklists are only modestly predictive of relapse so they could be improved by including more specific psychopathology.

Evidence suggests that 'basic symptoms' may be useful relapse indicators that could be added to checklists of conventional early warning signs to improve predictive power. Studies in individuals at high risk of psychosis have characterised basic symptoms as subtle, sub-clinical, qualitative disturbances in one's experience of oneself and the world which are predictive of transition to first episode psychosis. Typical basic symptoms include: changes in perceptions, such as increased vividness of colour vision; mild subjective cognitive problems; impaired tolerance to certain stressors; subjective difficulty finding or understanding common words. Two retrospective studies examining service users' experiences in the run up to a recent relapse of psychosis provide preliminary evidence that basic symptoms occur prior to relapse.

AIMS

The long term aim is to conduct a definitive study to prospectively investigate the predictive value of basic symptoms as early signs of psychosis relapse using a mobile phone application to monitor these within individuals' everyday lives. In line with the Medical Research Council guide for developing complex interventions a feasibility study will be conducted first. This study has four phases. In Phase 1 the investigators will design a measure of basic symptoms, assessed via smart-phone, and adapt it as applicable following feedback from participants. Phase 2 begins with a screening interview to identify participants with at least one basic symptom; these individuals will be eligible for Phase 3 (since past basic symptoms are likely to predict future basic symptoms). Cross-sectional assessments will also be conducted in Phase 2; by comparing those with and without basic symptoms the investigators will begin to characterise the sub-group of individuals with whom the basic symptom assessment can be used. In Phase 3 a prospective, longitudinal design will be used to investigate the feasibility of using a mobile phone application to regularly measure basic symptoms, conventional early signs and relapse over an extended period. Finally, in Phase 4, participants' experiences of using the phone application will be explored using qualitative interviews (acceptability).

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* current contact with mental health services
* a current, primary clinical diagnosis of non-affective psychotic disorder (DSM-IV)
* at least one episode of acute psychosis in the past year (admission to crisis team or hospital; or exacerbation of psychotic symptoms lasting at least 2 weeks and leading to a change in management), or at least two episodes of psychosis in the past 2 years, including index episode
* currently prescribed antipsychotic medication
* fluency in English
* fixed abode
* informed consent.

Exclusion Criteria:

* not sufficiently stable to take part (unable to complete screening assessment)
* significant history of organic factors implicated in the aetiology of psychotic symptoms
* current alcohol or drug dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with a schizophrenia spectrum diagnosis who have experienced at least one episode within the past year (or at least two within the past year) were recruited from three NHS mental health trusts in the North West of England.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Percentage of weekly app assessments completed per person during 6 month followup period | 6 months
  This is used as an indicator of the feasibility of using an app for 6 months

SECONDARY OUTCOMES:
Percentage of participants completing at least 33% of weekly app assessments during the 6 month followup period (retention) | 6 months
  This is used as an indicator of the feasibility of using an app for 6 months
Relapse rate: a symptom increase (measured using five PANSS items: delusions, hallucinations, grandiosity, suspiciousness, thought disorder) for at least one week that resulted in a management change as reported in casenotes | 6 months
  Symptom increase criteria were: for remitted individuals, an increase to four or above or an increase of at least two points (whichever was higher) on any item; for non-remitted individuals with all baseline PANSS positive items <5, at least one item ≥5; for non-remitted individuals with at least one baseline PANSS positive item ≥5, an increase of at least one point on any item. Individuals' initial remission status was determined from baseline PANSS interview using standard criteria. Remission status was updated during follow-up, based on app-assessed symptoms, using a parallel of the standard remission criteria (decrease to 3 or below on all app-assessed psychotic symptoms, for two consecutive weeks).
Selected items from the Basic Symptoms Checklist | Weekly for 6 months
  Weekly basic symptoms, assessed using items from the Basic Symptoms Checklist within the ExPRESS app
Selected items from the Early Signs Scale | Weekly for 6 months
  Weekly conventional early signs of relapse, assessed using items from the Early Signs Scale within the ExPRESS app
Selected items derived from the Positive and Negative Syndrome Scale (PANSS) | Weekly for 6 months
  Weekly psychotic symptoms, assessed using items derived from the Positive and Negative Syndrome Scale, within the ExPRESS app
Qualitative data from participant interviews regarding their experiences of using the ExPRESS app for 6 months | 6 months
  This is an indicator of acceptability of using an app for 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Emily Eisner, BA, MRes, Principal Investigator — University of Manchester

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Eisner E, Drake R, Lobban F, Bucci S, Emsley R, Barrowclough C. Comparing early signs and basic symptoms as methods for predicting psychotic relapse in clinical practice. Schizophr Res. 2018 Feb;192:124-130. doi: 10.1016/j.schres.2017.04.050. Epub 2017 May 9. PMID 28499766
- [Background] Eisner E, Drake R, Barrowclough C. Assessing early signs of relapse in psychosis: review and future directions. Clin Psychol Rev. 2013 Jul;33(5):637-53. doi: 10.1016/j.cpr.2013.04.001. Epub 2013 Apr 11. PMID 23628908
- [Background] Eisner E, Barrowclough C, Lobban F, Drake R. Qualitative investigation of targets for and barriers to interventions to prevent psychosis relapse. BMC Psychiatry. 2014 Jul 16;14:201. doi: 10.1186/1471-244X-14-201. PMID 25030092
- [Background] Robinson D, Woerner MG, Alvir JM, Bilder R, Goldman R, Geisler S, Koreen A, Sheitman B, Chakos M, Mayerhoff D, Lieberman JA. Predictors of relapse following response from a first episode of schizophrenia or schizoaffective disorder. Arch Gen Psychiatry. 1999 Mar;56(3):241-7. doi: 10.1001/archpsyc.56.3.241. PMID 10078501
- [Background] Appleby L. Suicide in psychiatric patients: risk and prevention. Br J Psychiatry. 1992 Dec;161:749-58. doi: 10.1192/bjp.161.6.749. PMID 1483160
- [Background] Wiersma D, Nienhuis FJ, Slooff CJ, Giel R. Natural course of schizophrenic disorders: a 15-year followup of a Dutch incidence cohort. Schizophr Bull. 1998;24(1):75-85. doi: 10.1093/oxfordjournals.schbul.a033315. PMID 9502547
- [Background] Mangalore R, Knapp M. Cost of schizophrenia in England. J Ment Health Policy Econ. 2007 Mar;10(1):23-41. PMID 17417045
- [Background] Almond S, Knapp M, Francois C, Toumi M, Brugha T. Relapse in schizophrenia: costs, clinical outcomes and quality of life. Br J Psychiatry. 2004 Apr;184:346-51. doi: 10.1192/bjp.184.4.346. PMID 15056580
- [Background] Herz MI, Lamberti JS, Mintz J, Scott R, O'Dell SP, McCartan L, Nix G. A program for relapse prevention in schizophrenia: a controlled study. Arch Gen Psychiatry. 2000 Mar;57(3):277-83. doi: 10.1001/archpsyc.57.3.277. PMID 10711914
- [Background] Lee SH, Choi TK, Suh S, Kim YW, Kim B, Lee E, Yook KH. Effectiveness of a psychosocial intervention for relapse prevention in patients with schizophrenia receiving risperidone via long-acting injection. Psychiatry Res. 2010 Feb 28;175(3):195-9. doi: 10.1016/j.psychres.2008.06.043. PMID 20022120
- [Background] Gumley A, O'Grady M, McNay L, Reilly J, Power K, Norrie J. Early intervention for relapse in schizophrenia: results of a 12-month randomized controlled trial of cognitive behavioural therapy. Psychol Med. 2003 Apr;33(3):419-31. doi: 10.1017/s0033291703007323. PMID 12701663
- [Background] Birchwood M, Smith J, Macmillan F, Hogg B, Prasad R, Harvey C, Bering S. Predicting relapse in schizophrenia: the development and implementation of an early signs monitoring system using patients and families as observers, a preliminary investigation. Psychol Med. 1989 Aug;19(3):649-56. doi: 10.1017/s0033291700024247. PMID 2798634
- [Background] Gumley AI, MacBeth A, Reilly JD, O'Grady M, White RG, McLeod H, Schwannauer M, Power KG. Fear of recurrence: results of a randomized trial of relapse detection in schizophrenia. Br J Clin Psychol. 2015 Mar;54(1):49-62. doi: 10.1111/bjc.12060. Epub 2014 Jul 8. PMID 25040487
- [Background] Norman RM, Malla AK. Prodromal symptoms of relapse in schizophrenia: a review. Schizophr Bull. 1995;21(4):527-39. doi: 10.1093/schbul/21.4.527. PMID 8749881
- [Background] Fusar-Poli P, Bonoldi I, Yung AR, Borgwardt S, Kempton MJ, Valmaggia L, Barale F, Caverzasi E, McGuire P. Predicting psychosis: meta-analysis of transition outcomes in individuals at high clinical risk. Arch Gen Psychiatry. 2012 Mar;69(3):220-9. doi: 10.1001/archgenpsychiatry.2011.1472. PMID 22393215
- [Background] Bechdolf A, Schultze-Lutter F, Klosterkotter J. Self-experienced vulnerability, prodromal symptoms and coping strategies preceding schizophrenic and depressive relapses. Eur Psychiatry. 2002 Nov;17(7):384-93. doi: 10.1016/s0924-9338(02)00698-3. PMID 12547304
- [Derived] Eisner E, Drake RJ, Berry N, Barrowclough C, Emsley R, Machin M, Bucci S. Development and Long-Term Acceptability of ExPRESS, a Mobile Phone App to Monitor Basic Symptoms and Early Signs of Psychosis Relapse. JMIR Mhealth Uhealth. 2019 Mar 29;7(3):e11568. doi: 10.2196/11568. PMID 30924789

DOCUMENTS (1):
  • Study Protocol (2016-08-26): https://cdn.clinicaltrials.gov/large-docs/29/NCT03558529/Prot_000.pdf